CLINICAL TRIAL: NCT03454230
Title: Pilot Study for Evaluation of the Procedure Impact of Mobilization Adapted to Pressure Ulcer Risk for Patients in Intensive Care.
Acronym: PROMESReaPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: K171008J; 2017-A03038-45 (Other: ANSM)
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pressure Ulcers; Nursing Cares; Decubitus Ulcer; Pressure Injury
Keywords: Intensive care unit; ICU; adult critical care patients; repositioning schedule; patient handling; practical nursing; nursing care; pressure ulcers; decubitus ulcers; pressure injury
MeSH Terms: conditions — Pressure Ulcer | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: To assess efficacy of a positioning schedule whose frequency of positioning is adapted every day to pressure ulcer risk assessed by Braden scale on occurrence of pressure ulcer in adult ICU in comparison with the routine patient management (without positioning schedule adapted on PU risk) at the 28th day, or when leaving ICU wall, or at death if it occurs before.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positioning schedule (Experimental): Applying repositioning schedule daily adapted to pressure ulcer risk assessed with Braden scale. Then, the nurse will applied oil for PU prevention and repositioning which frequency will be defined by the Braden score. The positions will be the semi-fowler 30-30, the half-sitting position with a 45° angle position and patient lying on their back with the head up with a 30° angle for ventilator associated pneumonia prevention.
  Repositioning schedule will be applied according to the daily medical prescription. When physician allows to sit the patient on a chair, this have to be done by raising feet on a stool. Therefore, patients will stay in that chair as long as defined by positioning schedule. When patient is returned to bed, same positions as described above will be used alternately. In the time of positioning care, oil usually used for PU prevention will be applied on the skin of the areas of high risk of PU (heels, sacrum, elbows, trochanter, knees) and bone projections.
  Interventions: Procedure: Positioning schedule
- Common repositioning practice (No Intervention): pressure ulcer prevention cares are provided according to usual practice. Frequency and modality of positioning applied to the patients are collected.

INTERVENTIONS:
Procedure: Positioning schedule — Applying repositioning schedule daily adapted to pressure ulcer risk assessed with Braden scale. Then, the nurse will applied oil for PU prevention and repositioning which frequency will be defined by the Braden score. The positions will be the semi-fowler 30-30, the half-sitting position with a 45° angle position and patient lying on their back with the head up with a 30° angle for ventilator associated pneumonia prevention.
  Repositioning schedule will be applied according to the daily medical prescription. When physician allows to sit the patient on a chair, this have to be done by raising feet on a stool. Therefore, patients will stay in that chair as long as defined by positioning schedule. When patient is returned to bed, same positions as described above will be used alternately. In the time of positioning care, oil usually used for PU prevention will be applied on the skin of the areas of high risk of PU (heels, sacrum, elbows, trochanter, knees) and bone projections.
  Other Names: Positioning; prevention of pressure ulcers; repositioning program
  Arms: Positioning schedule

SUMMARY:
Pressure ulcers (PU) represent a major health issue because of their high incidence and of their important consequences. There is an important risk of pressure ulcer acquisition for ICU patient with acute organ failure.

Specific risk factors identified in ICU are immobility, which accentuates the effects of friction and shears, as well as mechanical ventilation and the use of vasopressors.

A repositioning schedule is a guideline for pressure ulcer prevention, but repositioning frequency remains unknown.

Adaptation of the repositioning schedule to pressure ulcer risk assessment using Braden scale should decrease emergence of pressure ulcer. This could limit their important consequences for ICU patients which add to their brittle clinical condition (infection, increased length of stay, mortality…).

DETAILED DESCRIPTION:
This study will assess feasibility, efficacy and tolerance of a repositioning schedule applied to ICU adult patients. The repositioning schedule will be daily adapted to pressure ulcer risk of the patient assessed with Braden scale.

If results of this pilot study show improvement by the application of the repositioning schedule, they will argue the realization of a multicenter randomized clinical trial. This larger study will assess the expected decrease of pressure ulcers incidence due to the schedule and of its benefit-risk ratio.

This is a one-center prospective pilot study which includes two one-month consequential periods:

* During the first period, care will be delivered according usual practice. It is an observational phase.
* The second period will begin with medical and nurse staff training. Then, care will be delivered according the repositioning schedule. It's an interventional phase.

The procedure will be prescribed every day on patient's prescription by the doctor in charge (that will be filed with medical record).

- During the two periods: Every morning, inclusion and non-inclusion criteria will be sought for every patient intubated for at least 24 hours. This evaluation will be made by a nurse during daily medical staff meeting.

Eligible patients will be informed. Their consent will be collected and they will be included in the study. Patient characteristics (age, gender, BMI, simplified acute physiology score SAPS II, Sequential Organ Failure Assessment (SOFA) Score, length of mechanical ventilation, length of stay and mortality in ICU) will be taken from the PMSI. Those data are usually daily collected.

During the second period: data about Braden scale, positioning schedule, different positions applied, possible adverse events during positioning and presence of pressure ulcer will be collected by caregivers and nurses caring the patient.

Those data will be collected on the "daily positioning sheet" made available in patient's room. Skin condition will be evaluated on the 28th day, or when leaving ICU wall, or at death if it occurs before. Clinical research technician will control concordance between repositioning data and position applied by caregivers and nurses and those recommended by the schedule.

ELIGIBILITY:
Inclusion Criteria:

* Expected duration of invasive ventilation: more than 24 hours at inclusion;
* No pressure ulcer at inclusion (using of a tool developed from the European Pressure Ulcer Advisory Panel);;
* Information of the patient, or if it is not possible information of his relatives, or emergency procedure if contacting relatives is not possible. Consent document will then be signed by the patient as soon as he is able to do.

Exclusion Criteria:

* Under than 18 years;
* Pregnant woman;
* protected adult as defined by the law;
* Person without any health insurance;
* patient recruited in any other interventional research studying mobilization or positioning of the patient and/or pressure ulcer prevention and/or being in exclusion period of any other research if concerned;
* patient admitted in ICU for the multiple trauma management;
* patient concerned by a medical decision to limit active therapies at the time of potential inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
positioning schedule efficacy | 28 days
  To assess efficacy of a positioning schedule whose frequency of positioning is adapted every day to pressure ulcer risk assessed by Braden scale in adult ICU, compared to usual PU prevention management (without schedule daily adapted to PU risk) at the 28th day, or when leaving ICU wall, or at death if it occurs before.

SECONDARY OUTCOMES:
Caregivers commitment to the standardized positioning schedule in adult ICU (1) | 28 days
  Nurses commitment will be evaluated by accordance between frequency of positioning (mobilization frequency per day) according to the schedule and the frequency of positioning actually carried out by caregivers,
  These data will be collected by nurses on the "daily positioning sheet" made available in patient's room.
Caregivers commitment to the standardized positioning schedule in adult ICU (2) | 28 days
  Nurses commitment will be evaluated, by accordance between the positions planned by the schedule (Right Semi-Lateral Decubitus, Left Semi-Lateral Decubitus, Semi-Fowler 30 °, Half-Seated 45 °, Seated in Armchair) and those actually achieved by caregivers.
  These data will be collected by nurses on the "daily positioning sheet" made available in patient's room.
nursing workload | 28 days
  To assess the workload added to nursing care by the positioning schedule : nursing workload will be assessed by the total time dedicated for positioning the patient. This time will be calculated in minutes, from positioning time notified on the "daily positioning sheet". It will be reported on the "positioning sheet stay" by the clinical research technician.
clinical safety of the positioning schedule | 28 days
  To assess the clinical safety of the positioning schedule : the clinical safety will be assessed by the percentage of adverse events occurrence during when positioning the patients.
  Adverse events are defined as accidental removal of invasive devices (breathing tube, catheter, chest tube, gastric tube, urinary catheter) and an instability (hemodynamic or respiratory) requiring positioning discontinuation. Caregivers monitor vital parameters during positioning and discontinue the positioning if hemodynamic or respiratory instability occurs, according to nurse's clinical evaluation. Adverse events will be notified on the "daily positioning sheet" and on the "positioning sheet stay" by caregivers charge positioning the patient.

CONTACTS AND LOCATIONS:
Overall Officials: MEHAY Daisy, RN, Principal Investigator — Service de réanimation médico chirurgicale, Hôpital Tenon (AP-HP), Paris; FARTOUKH Muriel, MD, Study Director — Service de réanimation médico chirurgicale, Hôpital Tenon (AP-HP), Paris
Locations (1):
- Hôpital Tenon, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No
It is planned to share data to argue the realization of a multicenter trial on this theme. This data can be shared by different way including e-mail transfer.